CLINICAL TRIAL: NCT02422264
Title: Immunogenicity and Safety Study of GSK Biologicals' Combined Diphtheria-tetanus-acellular Pertussis-hepatitis B-inactivated Polio-virus and Haemophilus Influenzae Type b Vaccine (Infanrix Hexa™) (217744) in Healthy Infants Born to Mothers Vaccinated With Boostrix™ During Pregnancy or Immediately Post-delivery
Brief Title: Immunogenicity and Safety Study of Infanrix Hexa in Healthy Infants Born to Mothers Vaccinated With Boostrix™ During Pregnancy or Immediately Post-delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201330; 2014-001117-41 (EudraCT Number)
Record Dates: First submitted 2015-03-19; First posted 2015-04-21 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Acellular Pertussis; Tetanus; Poliomyelitis; Diphtheria; Diphtheria-Tetanus-aPertussis-Hepatitis B-Poliomyelitis-Haemophilus Influenzae Type b Vaccines
MeSH Terms: conditions — Tetanus; Poliomyelitis; Diphtheria | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No

ARMS (2):
- dTpa Group (Experimental): This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047] i.e. who received a single dose of BoostrixTM during pregnancy and a dose of placebo immediately post-delivery. All infants in this group will receive Infanrix hexaTM co-administered with Prevenar 13®.
  Interventions: Biological: Infanrix hexa; Drug: Prevnar13
- Control Group (Active Comparator): This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047], i.e. who received a single dose of placebo during pregnancy and a dose of BoostrixTM immediately post-delivery. All infants in this group will receive Infanrix hexaTM co-administered with Prevenar 13®.
  Interventions: Biological: Infanrix hexa; Drug: Prevnar13

INTERVENTIONS:
Biological: Infanrix hexa — • All subjects will receive Infanrix hexa at 2 and 4, at 3 and 5, at 2, 4 and 6 months or at 2, 3 and 4 months, depending on the immunisation schedule of the country. Infanrix hexa is administered intramuscularly to the right thigh.
Drug: Prevnar13 — • All subjects will receive Infanrix hexa co-administered with Prevenar13* at 2 and 4, at 3 and 5, at 2, 4 and 6 months or at 2, 3 and 4 months, depending on the immunisation schedule of the country. *In some countries/regions with an Infanrix hexa 3-dose vaccination schedule, Prevenar 13 could be administered as 2-doses or 3-doses primary vaccination schedule (according to the routine national immunisation schedule). Prevnar13 is administered intramuscularly to the left thigh.

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of GSK Biologicals' Infanrix hexa, given in the primary vaccination schedule to infants born to pregnant women who participated in study 116945 [DTPA (BOOSTRIX)-047]. This study will help us evaluate if the presence of transplacentally transferred maternal antibodies interfere with the immune response to primary vaccination with Infanrix hexa and a co-administered pneumococcal conjugate vaccine given as a part of this study in infants.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply, with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits).
* Written informed consent obtained from the parent(s)/LAR(s) of the subject prior to performing any study specific procedure.
* A male or female between, 6 and 14 weeks of age (including 6 weeks and up to and including 14 weeks and 6 days of age) at the time of the first vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born to a mother enrolled in study 116945 [DTPA (BOOSTRIX)-047].
* Medically stable* prematurely born infants, born after a gestation period of 27-36 weeks may be enrolled in the study at the discretion of the investigator.

  * Medically stable refers to the condition of premature infants who do not require significant medical support or ongoing management for debilitating disease and who have demonstrated a clinical course of sustained recovery by the time they receive the first dose of study vaccine.

Exclusion Criteria:

* Child in care
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting at birth prior to the first vaccine dose. For corticosteroids, this will mean prednisone ≥0.5mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
* Administration of any chronic drug therapy to be continued during the study period.
* A vaccine not foreseen by the study protocol administered during the period starting from 30 days before each dose of vaccine and ending 30 days after*, with the exception of inactivated influenza vaccine and other vaccines given as a part of the national/regional immunisation schedule, that are allowed at any time during the study period.

  * In case an emergency mass vaccination for an unforeseen public health threat (e.g.: a pandemic) is organised by the public health authorities, outside the routine immunisation program, the time period described above can be reduced if necessary for that vaccine provided it is licensed and used according to its SPC or package insert (PI) and according to the local governmental recommendations and provided a written approval of the Sponsor is obtained.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Previous vaccination against Hib, diphtheria, tetanus, pertussis, pneumococcus, and/or poliovirus since birth.
* History of Hib, diphtheria, tetanus, pertussis, pneumococcal, poliovirus and hepatitis B diseases.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including severe combined immunodeficiency disease (SCID), based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Major congenital defects
* Serious chronic illness.
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥37.5°C/99.5°F for oral, axillary or tympanic route, or ≥38.0°C/100.4°F for rectal route.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products during the period starting at birth before the first dose of study vaccines or planned administration during the study period.
* Hypersensitivity to latex.

Ages: 6 Weeks to 14 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 601 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- GSK Investigational Site, Carlton, Victoria, Australia
- Canada (3):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Montreal, Quebec
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Ostrava - Vitkovice
  - GSK Investigational Site, Prague
- Finland (5):
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Italy (3):
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Novara, Piedmont
  - GSK Investigational Site, Turin, Piedmont
- Spain (9):
  - GSK Investigational Site, Málaga, Andalusia
  - GSK Investigational Site, Antequera/Málaga
  - GSK Investigational Site, Aravaca
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Móstoles
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Perrett KP, Halperin SA, Nolan T, Carmona Martinez A, Martinon-Torres F, Garcia-Sicilia J, Virta M, Vanderkooi OG, Zuccotti GV, Manzoni P, Kostanyan L, Meyer N, Ceregido MA, Cheuvart B, Kuriyakose SO, Stranak Z, Merino Arribas JM, Cilleruelo Ortega MJ, Miranda-Valdivieso M, Arias Novas B, Ramos Amador JT, Omenaca F, Baca M, Marchisio PG, Mesaros N. Impact of tetanus-diphtheria-acellular pertussis immunization during pregnancy on subsequent infant immunization seroresponses: follow-up from a large randomized placebo-controlled trial. Vaccine. 2020 Feb 18;38(8):2105-2114. doi: 10.1016/j.vaccine.2019.10.104. Epub 2019 Nov 24. PMID 31776027

RESULTS

PARTICIPANT FLOW:
Groups:
- dTpa Group: Infants born to mothers belonging to the Boostrix Group in study NCT02377349 [DTPA (BOOSTRIX)-047] i.e. who received a single dose of Boostrix during pregnancy and a dose of placebo immediately post-delivery. All infants in this group received Infanrix hexa co-administered with Prevenar 13 according to the routine national immunisation schedule.
- Control Group: Infants born to mothers belonging to the Control group in study NCT02377349 [DTPA (BOOSTRIX)-047], i.e. who received a single dose of placebo during pregnancy and a dose of Boostrix immediately post-delivery. All infants in this group received Infanrix hexa co-administered with Prevenar 13 according to the routine national immunisation schedule.
Period: Overall Study
Arm/Group | dTpa Group | Control Group
Started | 296 | 305
Completed | 291 | 301
Not Completed | 5 | 4
Not completed — Serious Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Migrated/moved from study area | 3 | 1
Not completed — Subject vaccinated outside of the study | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | dTpa Group | Control Group | Total
Number analyzed (Participants) | 296 | 305 | 601
Age, Continuous [Mean (Standard Deviation); unit: Weeks] — Age at Dose 1
  Weeks | 8.7 (1.6) | 8.9 (1.8) | 8.8 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 144 | 285
  Male | 155 | 161 | 316
Race/Ethnicity, Customized [Number; unit: Participants]
  African Heritage / African American | 4 | 9 | 13
  Asian - East Asian Heritage | 2 | 0 | 2
  Asian - South East Asian Heritage | 3 | 0 | 3
  White - Arabic / North African Heritage | 1 | 3 | 4
  White - Caucasian / European Heritage | 268 | 285 | 553
  Mixed origin | 18 | 8 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Vaccine Response Against Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN) Antigens
Description: Vaccine response to the PT, FHA and PRN antigens, is defined as the appearance of antibodies in subjects who were initially seronegative (i.e., with concentrations lower than (<) the cut-off value of the assay), or at least maintenance of pre-vaccination antibody concentrations in subjects who were initially seropositive (i.e., with concentrations greater than or equal to (≥) the cut-off value of the assay). Assay cut-off was 2.693 IU/mL for anti-PT, 2.046 IU/mL for anti-FHA, 2.187 IU/mL for anti-PRN.
Time Frame: 1 month after the last dose of the primary vaccination
Population: The analysis was performed on the According to Protocol (ATP) cohort for immunogenicity, which included all subjects from the Totally vaccinated cohort (TVC) who complied with the vaccine administration and with the protocol and for whom data concerning immunogenicity outcome measures were available for at least one study vaccines antigen component
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 240 | 251
Participants
  anti-PT antibody | 185 | 249
  anti-FHA antibody | 95 | 238
  anti-PRN antibody: number analyzed (Participants) | 240 | 250
  anti-PRN antibody | 90 | 225

2. Primary Outcome: Number of Seroprotected Subjects With Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibody Concentration Above or Equal to the Assay Cut-off
Description: A seroprotected subject is a subject whose antibody concentration/titre was ≥ the level defining clinical protection, of 0.1 International Units per milliliter (IU/mL).
Time Frame: 1 month after the last dose of the primary vaccination
Population: The analysis was performed on the According to Protocol (ATP) cohort for immunogenicity, which included all subjects from the TVC who complied with the vaccine administration and with the protocol and for whom data concerning immunogenicity outcome measures were available for at least one study vaccines antigen component.
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 266 | 271
Participants
  anti-D antibody: number analyzed (Participants) | 264 | 271
  anti-D antibody | 264 | 271
  anti-T antibody | 266 | 271

3. Primary Outcome: Number of Seroprotected Subjects With Anti Hepatitis B (Anti-HBs) Antibody Concentration Above or Equal to the Assay Cut-off
Description: A seroprotected subject is a subject whose antibody concentration/titre was ≥ to the level defining clinical protection, of 10 micro International Units per milliliter (mIU/mL).
Time Frame: 1 month after the last dose of the primary vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 253 | 263
Participants | 251 | 259

4. Primary Outcome: Number of Seroprotected Subjects With Anti-poliovirus Type 1, 2 and 3 Antibody Concentration Above or Equal to 8
Description: A seroprotected subject is a subject whose antibody titre was ≥ the level defining clinical protection, of 8 ED50.
Time Frame: 1 month after the last dose of the primary vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 241 | 245
Participants
  anti-Polio 1 antibody: number analyzed (Participants) | 237 | 244
  anti-Polio 1 antibody | 233 | 242
  anti-Polio 2 antibody | 239 | 235
  anti-Polio 3 antibody: number analyzed (Participants) | 230 | 237
  anti-Polio 3 antibody | 228 | 236

5. Primary Outcome: Number of Seroprotected Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentration Above or Equal to the Assay Cut-off
Description: A seroprotected subject is a subject whose antibody concentration/titre was ≥ the level defining clinical protection, of 0.15 micrograms per milliliter (µg/mL).
Time Frame: 1 month after the last dose of the primary vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 266 | 271
Participants | 255 | 256

6. Secondary Outcome: Number of Seroprotected Subjects Against Diphtheria (Anti-D) and Tetanus (Anti-T) Antibody Concentration Above or Equal to the Assay Cut-off.
Description: A seroprotected subject is a subject whose antibody concentration was ≥ the level defining clinical protection, of 0.1 IU/mL.
Time Frame: Before the first dose of Infanrix hexa
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 242 | 253
Participants
  anti-D antibody: number analyzed (Participants) | 242 | 252
  anti-D antibody | 200 | 110
  anti-T antibody | 240 | 225

7. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Antibody concentrations were expressed as geometric mean concentrations (GMCs) and measured in IU/mL.
Time Frame: Before the first dose of Infanrix hexa
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 242 | 253
IU/mL
  anti-D antibody: number analyzed (Participants) | 242 | 252
  anti-D antibody | 0.423 [0.354 to 0.506] | 0.089 [0.076 to 0.103]
  anti-T antibody | 2.152 [1.925 to 2.406] | 0.378 [0.330 to 0.434]

8. Secondary Outcome: Number of Subjects With Anti-PT, Anti-FHA and Anti-PRN Antibody Concentration Above or Equal to the Assay Cut-off.
Description: A seropositive subject is a subject whose antibody concentration is ≥ the assay cut-off defined. Assay cut-off was 2.693 IU/mL for anti-PT, 2.046 IU/mL for anti-FHA,2.187 IU/mL for anti-PRN
Time Frame: Before the first dose of Infanrix hexa
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 242 | 253
Participants
  anti-PT antibody | 218 | 88
  anti-FHA antibody | 242 | 210
  anti-PRN antibody | 231 | 151

9. Secondary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Anti-PT, anti-FHA and anti-PRN antibody concentrations were expressed as GMCs and measured in IU/mL.
Time Frame: Before the first dose of Infanrix hexa
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 242 | 253
IU/ml
  anti-PT antibody | 11.9 [10.3 to 13.6] | 2.2 [2.0 to 2.5]
  anti-FHA antibody | 88.3 [77.7 to 100.4] | 6.6 [5.7 to 7.7]
  anti-PRN antibody | 70.5 [56.1 to 88.5] | 4.5 [3.7 to 5.4]

10. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Antibody concentrations were expressed as geometric mean concentrations (GMCs) and measured in IU/mL.
Time Frame: 1 month after the last dose of the primary vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 266 | 271
IU/ml
  anti-D antibody: number analyzed (Participants) | 264 | 271
  anti-D antibody | 1.747 [1.598 to 1.910] | 2.746 [2.502 to 3.015]
  anti-T antibody | 2.347 [2.135 to 2.582] | 2.278 [2.069 to 2.508]

11. Secondary Outcome: Anti-Polio Type 1, 2 and 3 Antibody Titers
Description: Anti-Polio type 1, 2 and 3 antibody titers were expressed as geometric mean titers (GMT).
Time Frame: 1 month after the last dose of the primary vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 241 | 245
Titers
  anti-Polio 1 antibody: number analyzed (Participants) | 237 | 244
  anti-Polio 1 antibody | 432.1 [351.8 to 530.9] | 489.9 [402.6 to 596.0]
  anti-Polio 2 antibody | 424.6 [342.7 to 526.2] | 388.4 [306.3 to 492.6]
  anti-Polio 3 antibody: number analyzed (Participants) | 230 | 237
  anti-Polio 3 antibody | 730.6 [596.5 to 894.9] | 775.6 [645.9 to 931.3]

12. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Anti-HBs antibody concentrations were expressed as geometric mean concentrations (GMCs) and measured in mIU/mL.
Time Frame: 1 month after the last dose of the primary vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/ml
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 253 | 263
mIU/ml | 1322.8 [1116.7 to 1567.0] | 1339.2 [1132.8 to 1583.3]

13. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Anti-PRP antibody concentrations were expressed as GMCs and measured in µg/mL.
Time Frame: 1 month after the last dose of the primary vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 266 | 271
µg/mL | 1.862 [1.554 to 2.231] | 1.717 [1.428 to 2.064]

14. Secondary Outcome: Anti-PT, Anti-FHA, Anti-PRN Antibody Concentrations
Description: Anti-PT, anti-FHA, anti-PRN antibody concentrations were expressed as GMCs and measured in IU/mL.
Time Frame: 1 month after the last dose of the primary vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 266 | 271
IU/mL
  anti-PT antibody | 32.7 [30.2 to 35.3] | 54.7 [51.0 to 58.6]
  anti-FHA antibody | 68.5 [63.5 to 73.9] | 103.5 [95.6 to 112.1]
  anti-PRN antibody: number analyzed (Participants) | 266 | 270
  anti-PRN antibody | 60.5 [54.2 to 67.6] | 92.0 [81.6 to 103.6]

15. Secondary Outcome: Anti-pneumococcal Antibody Concentrations
Description: Assessed anti-pneumococcal serotypes were (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F), expressed as GMCs and measured in µg/mL.
Time Frame: 1 month after the last dose of the primary vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 232 | 237
µg/mL
  anti-PnPS 1 antibody | 1.61 [1.43 to 1.80] | 1.92 [1.73 to 2.14]
  anti-PnPS 3 antibody | 0.54 [0.49 to 0.60] | 0.60 [0.55 to 0.67]
  anti-PnPS 4 antibody | 1.20 [1.07 to 1.35] | 1.56 [1.40 to 1.75]
  anti-PnPS 5 antibody: number analyzed (Participants) | 226 | 234
  anti-PnPS 5 antibody | 1.09 [0.96 to 1.24] | 1.27 [1.13 to 1.43]
  anti-PnPS 6A antibody | 2.16 [1.89 to 2.47] | 2.59 [2.27 to 2.95]
  anti-PnPS 6B antibody | 1.37 [1.12 to 1.68] | 1.44 [1.20 to 1.73]
  anti-PnPS 7F antibody | 2.39 [2.15 to 2.65] | 2.67 [2.43 to 2.93]
  anti-PnPS 9V antibody | 1.33 [1.19 to 1.50] | 1.64 [1.47 to 1.83]
  anti-PnPS 14 antibody | 5.70 [4.99 to 6.52] | 6.57 [5.71 to 7.56]
  anti-PnPS 18C antibody | 1.61 [1.42 to 1.82] | 1.79 [1.59 to 2.01]
  anti-PnPS 19A antibody | 1.61 [1.43 to 1.82] | 2.01 [1.78 to 2.27]
  anti-PnPS 19F antibody | 2.57 [2.35 to 2.82] | 3.24 [2.92 to 3.60]
  anti-PnPS 23F antibody: number analyzed (Participants) | 230 | 236
  anti-PnPS 23F antibody | 0.86 [0.74 to 0.99] | 1.02 [0.88 to 1.17]

16. Secondary Outcome: Number of Subjects With Anti-PT, Anti-FHA, Anti-PRN Antibody Concentration Above or Equal to the Assay Cut-off.
Description: as for outcome 8
Time Frame: 1 month after the last dose of the primary vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 266 | 271
Participants
  anti-PT antibody | 266 | 271
  anti-FHA antibody | 266 | 271
  anti-PRN antibody: number analyzed (Participants) | 266 | 270
  anti-PRN antibody | 266 | 269

17. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Solicited local symptoms were assessed by each and across dose.
Time Frame: During the 4-day (Day 0-Day 3) follow-up period after each vaccination
Population: The analysis was performed on the Total vaccinated cohort (TVC), which included all vaccinated subjects for whom data were available and for those with at least 1 vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 294 | 303
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 293 | 301
  Any Pain, Dose 1 | 120 | 120
  Any Redness, Dose 1 | 128 | 116
  Any Swelling, Dose 1 | 81 | 87
  Any Pain, Dose 2: number analyzed (Participants) | 288 | 303
  Any Pain, Dose 2 | 109 | 101
  Any Redness, Dose 2: number analyzed (Participants) | 288 | 303
  Any Redness, Dose 2 | 139 | 139
  Any Swelling, Dose 2: number analyzed (Participants) | 288 | 303
  Any Swelling, Dose 2 | 98 | 95
  Any Pain, Dose 3: number analyzed (Participants) | 259 | 260
  Any Pain, Dose 3 | 85 | 94
  Any Redness, Dose 3: number analyzed (Participants) | 259 | 260
  Any Redness, Dose 3 | 122 | 134
  Any Swelling, Dose 3: number analyzed (Participants) | 259 | 260
  Any Swelling, Dose 3 | 77 | 109
  Any Pain, Across Doses | 175 | 184
  Any Redness, Across Doses | 205 | 203
  Any Swelling, Across Doses | 157 | 168

18. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability/fussiness, loss of appetite and fever [defined as axillary route temperature ≥ 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Solicited general symptoms were assessed by each and across dose.
Time Frame: During the 4-day (Day 0-Day 3) follow-up period after each vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 294 | 303
Participants
  Any Drowsiness, Dose 1: number analyzed (Participants) | 294 | 300
  Any Drowsiness, Dose 1 | 166 | 174
  Any Irritability / Fussiness, Dose 1: number analyzed (Participants) | 294 | 300
  Any Irritability / Fussiness, Dose 1 | 187 | 191
  Any Loss of Appetite, Dose 1: number analyzed (Participants) | 293 | 300
  Any Loss of Appetite, Dose 1 | 85 | 94
  Any Temperature/(Axillary) (≥37.5°C), Dose 1: number analyzed (Participants) | 293 | 300
  Any Temperature/(Axillary) (≥37.5°C), Dose 1 | 64 | 69
  Any Drowsiness, Dose 2: number analyzed (Participants) | 288 | 303
  Any Drowsiness, Dose 2 | 142 | 149
  Any Irritability / Fussiness, Dose 2: number analyzed (Participants) | 288 | 303
  Any Irritability / Fussiness, Dose 2 | 182 | 194
  Any Loss of Appetite, Dose 2: number analyzed (Participants) | 288 | 303
  Any Loss of Appetite, Dose 2 | 69 | 94
  Any Temperature/(Axillary) (≥37.5°C), Dose 2: number analyzed (Participants) | 288 | 303
  Any Temperature/(Axillary) (≥37.5°C), Dose 2 | 62 | 76
  Any Drowsiness, Dose 3: number analyzed (Participants) | 259 | 260
  Any Drowsiness, Dose 3 | 99 | 104
  Any Irritability / Fussiness, Dose 3: number analyzed (Participants) | 259 | 260
  Any Irritability / Fussiness, Dose 3 | 142 | 161
  Any Loss of Appetite, Dose 3: number analyzed (Participants) | 259 | 260
  Any Loss of Appetite, Dose 3 | 64 | 63
  Any Temperature/(Axillary) (≥37.5°C), Dose 3: number analyzed (Participants) | 259 | 260
  Any Temperature/(Axillary) (≥37.5°C), Dose 3 | 52 | 47
  Any Drowsiness, Across Doses | 216 | 232
  Any Irritability/Fussiness, Across Doses | 255 | 257
  Any Loss of appetite, Across Doses | 142 | 157
  Any Temperature/(Axillary) (≥37.5°C), Across Doses | 125 | 126

19. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any is defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (days 0-30) follow-up period after each vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 296 | 305
Participants | 161 | 173

20. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed included medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity.
Time Frame: From Day 0, prior to vaccination until the study end, at Month 3 or 5 (depending on vaccination schedule of the country)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 296 | 305
Participants | 7 | 17

ADVERSE EVENTS:
Time Frame: Solicited symptoms were collected during the 4-day (Day 0-Day 3) follow-up period after each vaccination. Unsolicited AEs were collected during the 31-day (days 0-30) follow-up period after each vaccination. SAEs were collected from Day 0 to Month 3 or 5.
Arm/Group | dTpa Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/296 | 0/305
Serious Adverse Events (participants affected / at risk) | 7/296 | 17/305
Other Adverse Events (participants affected / at risk) | 292/296 | 294/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | dTpa Group (N=296) | Control Group (N=305)
Congenital cytomegalovirus infection (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Craniosynostosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Dandy-walker syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ear malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Microcephaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Milk allergy (Immune system disorders) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 4 (5)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Superinfection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | dTpa Group (N=296) | Control Group (N=305)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Congenital torticollis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 2 (2)
Eye discharge (Eye disorders) | 0 (0) | 2 (2)
Eye irritation (Eye disorders) | 1 (1) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Pupils unequal (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (9) | 9 (10)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 2 (2)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (8) | 6 (6)
Gingival pain (Gastrointestinal disorders) | 4 (5) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Infantile colic (Gastrointestinal disorders) | 2 (2) | 2 (2)
Infrequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral mucosal erythema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sandifer's syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Teething (Gastrointestinal disorders) | 14 (21) | 14 (16)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 4 (4)
Influenza like illness (General disorders) | 3 (3) | 0 (0)
Injection site bruising (General disorders) | 2 (2) | 2 (2)
Injection site induration (General disorders) | 1 (1) | 0 (0)
Injection site mass (General disorders) | 3 (4) | 1 (2)
Injection site nodule (General disorders) | 1 (1) | 1 (1)
Injection site swelling (General disorders) | 157 (256) | 169 (292)
Pyrexia (General disorders) | 133 (203) | 139 (208)
Thirst (General disorders) | 1 (1) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 2 (2)
Vaccination site pain (General disorders) | 1 (1) | 0 (0)
Vaccination site swelling (General disorders) | 1 (1) | 1 (1)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1)
Milk allergy (Immune system disorders) | 1 (1) | 2 (2)
Adenoiditis (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 5 (5) | 11 (12)
Bronchitis (Infections and infestations) | 4 (4) | 5 (6)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 2 (2) | 0 (0)
Candida nappy rash (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 6 (6) | 13 (14)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 6 (6) | 10 (12)
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Erythema infectiosum (Infections and infestations) | 1 (1) | 0 (0)
Exanthema subitum (Infections and infestations) | 1 (1) | 3 (3)
Eye infection (Infections and infestations) | 1 (2) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 5 (5) | 8 (8)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 2 (2)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 3 (3) | 3 (3)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 20 (21) | 15 (17)
Oral candidiasis (Infections and infestations) | 4 (4) | 2 (2)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 3 (3)
Otitis media acute (Infections and infestations) | 3 (3) | 2 (3)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 4 (5) | 9 (12)
Respiratory tract infection viral (Infections and infestations) | 4 (4) | 8 (8)
Rhinitis (Infections and infestations) | 2 (2) | 8 (8)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 36 (41) | 32 (38)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Body temperature increased (Investigations) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 142 (219) | 157 (252)
Head deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Positional plagiocephaly (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Infantile haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1)
External hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 2 (2) | 3 (3)
Genital labial adhesions (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 13 (14)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 8 (8)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (7)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 9 (9)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 205 (389) | 203 (389)
Injection site pain (General disorders) | 175 (314) | 184 (315)
Irritability postvaccinal (General disorders) | 255 (511) | 257 (546)
Somnolence (Nervous system disorders) | 216 (407) | 232 (427)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-09-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT02422264/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT02422264/SAP_001.pdf